CLINICAL TRIAL: NCT00778258
Title: Dietary Intervention in Milk Allergy and Tolerance Development
Brief Title: Study of Milk Allergy and Tolerance in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Asthma and Allergic Diseases Cooperative Research Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT AADCRC-MSSM-02
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Food Hypersensitivity; Milk Hypersensitivity
Keywords: Food Allergy; Milk Allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Milk-allergic; Non-consumption (Experimental): Subjects in this arm reacted to the lowest baseline dose of baked milk (muffin) and will continue strict milk avoidance, returning for re-evaluation with laboratory tests at 12 and 24 months and baked milk challenge at 36 months. Individual participants may be challenged at 12 and or 24 months.
  Interventions: Biological: Baked Milk
- Tolerated Muffin, Reacted to Pizza (Experimental): Subjects will be assigned to this arm, if they can tolerate ingesting a muffin but react to ingesting the amount of baked milk in a standardized portion of pizza. Within the arm, subjects will be randomized in 1:1 ratio to either return for re-evaluation at 6 months (Dose Escalation sub-arm) or 12 months (Maintenance sub-arm) to determine whether they might progress to ingesting higher amounts of baked milk protein.
  Interventions: Biological: Baked Milk
- Reacted to Rice Pudding (Experimental): Subjects will be assigned to this arm, if they can tolerate ingesting a muffin and a standardized portion of pizza but react to a standardized dose of baked milk in rice pudding. Within the arm, subjects will be randomized in 1:1 ratio to either return for re-evaluation at 6 months (Dose Escalation sub-arm) or 12 months (Maintenance sub-arm) to determine whether they might progress to ingesting higher amounts of baked milk protein.
  Interventions: Biological: Baked Milk
- Reacted to Non-baked Milk (Experimental): Subjects will be assigned to this arm, if they can tolerate ingesting a muffin, pizza and rice pudding but react to a standardized dose of non-baked milk. Within the arm, subjects will be randomized in 1:1 ratio to either return for re-evaluation at 6 months (Dose Escalation sub-arm) or 12 months (Maintenance sub-arm) to determine whether they might progress to ingesting higher amounts of baked milk protein.
  Interventions: Biological: Baked Milk; Biological: Non-baked Milk
- Tolerant to Baked and Non-baked Milk (Experimental): Biological/Vaccine: Baked Milk At baseline, each subject will undergo sequential oral food challenges with the products that contain increasing amounts of milk protein that are baked: Stage 1 (muffin), Stage 2 (pizza), and Stage 3 (rice pudding) doses of baked milk to determine the extent to which they tolerate various baked milk proteins. Based on the outcomes of the baseline oral food challenges, subjects will be assigned to one of the 5 study arms.
  Biological/Vaccine: Non-baked Milk Those subjects tolerant to rice pudding will undergo oral food challenge with non-baked milk.
  Interventions: Biological: Baked Milk; Biological: Non-baked Milk
- Non-Interventional Comparison (No Intervention): Thirty subjects who fulfill inclusion criteria but are unwilling to participate in the full protocol will be enrolled as a comparison group to the active arms.

INTERVENTIONS:
Biological: Baked Milk — At baseline, each subject will undergo sequential oral food challenges with the products that contain increasing amounts of milk protein that are baked: Stage 1 (muffin), Stage 2 (pizza), and Stage 3 (rice pudding) doses of baked milk to determine the extent to which they tolerate various baked milk proteins. Based on the outcomes of the baseline oral food challenges, subjects will be assigned to one of the 5 study arms.
  Arms: Milk-allergic; Non-consumption; Reacted to Non-baked Milk; Reacted to Rice Pudding; Tolerant to Baked and Non-baked Milk; Tolerated Muffin, Reacted to Pizza
Biological: Non-baked Milk — Those subjects tolerant to rice pudding will undergo oral food challenge with non-baked milk.
  Arms: Reacted to Non-baked Milk; Tolerant to Baked and Non-baked Milk

SUMMARY:
The purpose of this study is to determine if children who are allergic to milk can increase tolerance through frequent dose-escalation every 6 months versus 12 months leading to eventual tolerance of less heated milk and ultimately unheated milk.

DETAILED DESCRIPTION:
Milk is among the most common food allergens in infants and children. The majority of children outgrow their milk allergies; however, the exact mechanisms by which food tolerance is achieved are unknown. Strict avoidance of the offending food is currently the only known therapy. However, some have been known to tolerate milk products cooked at high heat such as when baked in foods.

This clinical trial involves a diet containing extensively baked milk protein to investigate the effects of ingestion of heat-denatured milk on development of oral tolerance to non-baked milk.

ELIGIBILITY:
Inclusion Criteria:

One or more of the following inclusion criteria for enrollment in the study have to be met:

* Convincing history of an allergic reaction to milk or a positive double blind placebo controlled milk challenge (DBPCMC) within the past 2 years and either detectable milk immunoglobulin E (IgE) or positive prick skin test to milk OR
* Serum milk-IgE of high predictive value >14 kUa/L or prick skin test to milk > 10mm wheal within the past 6 months regardless of past clinical history of reactions OR
* Convincing history of an allergic reaction to milk or a positive DBPCMC more than 2 years ago and either a positive serum milk-IgE < 14 kUA/L or positive prick skin test to milk < 10 mm wheal within the past 6 months (eligible only for the active arm of the study and will undergo a reversed sequence of initial baked-milk challenges)

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or to comply with study protocol

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2008-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A. Sampson, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Anna Nowak-Wegrzyn, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Nowak-Wegrzyn A, Bloom KA, Sicherer SH, Shreffler WG, Noone S, Wanich N, Sampson HA. Tolerance to extensively heated milk in children with cow's milk allergy. J Allergy Clin Immunol. 2008 Aug;122(2):342-7, 347.e1-2. doi: 10.1016/j.jaci.2008.05.043. Epub 2008 Jul 11. PMID 18620743
- [Background] Skripak JM, Matsui EC, Mudd K, Wood RA. The natural history of IgE-mediated cow's milk allergy. J Allergy Clin Immunol. 2007 Nov;120(5):1172-7. doi: 10.1016/j.jaci.2007.08.023. Epub 2007 Nov 1. PMID 17935766
- [Background] Staden U, Rolinck-Werninghaus C, Brewe F, Wahn U, Niggemann B, Beyer K. Specific oral tolerance induction in food allergy in children: efficacy and clinical patterns of reaction. Allergy. 2007 Nov;62(11):1261-9. doi: 10.1111/j.1398-9995.2007.01501.x. PMID 17919140
- [Background] Vandenplas Y, Koletzko S, Isolauri E, Hill D, Oranje AP, Brueton M, Staiano A, Dupont C. Guidelines for the diagnosis and management of cow's milk protein allergy in infants. Arch Dis Child. 2007 Oct;92(10):902-8. doi: 10.1136/adc.2006.110999. PMID 17895338
- See also: Description of NIAID Asthma and Allergic Diseases Cooperative Research Centers (AADCRC) Program — http://www.niaid.nih.gov/TOPICS/ASTHMA/RESEARCH/Pages/AADCRCs.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation - Reacted to Pizza: At baseline, participants had an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to pizza and were then randomized to return for re-evaluation every 6 months (dose escalation) to determine whether they might progress to ingesting higher amounts of baked milk protein. Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
- Dose Escalation - Reacted to Rice Pudding: At baseline, participants performed an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to rice pudding and were then randomized to return for re-evaluation every 6 months (dose escalation) to determine whether they might progress to ingesting higher amounts of baked milk protein. Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
- Dose Escalation - Reacted to Non-baked Milk: At baseline, participants performed an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to non-baked milk and were then randomized to re-try less denatured milk protein food items every 6 months (dose escalation). Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
- Maintenance - Reacted to Pizza: At baseline, participants had an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to pizza and were then randomized to return for re-evaluation every 12 months (maintenance) to determine whether they might progress to ingesting higher amounts of baked milk protein. Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
- Maintenance - Reacted to Rice Pudding; Maintenance- Reacted to Non-baked Milk: At baseline, participants had an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to rice pudding and were then randomized to continue eating the food at the same level of milk denaturalization and come in for OFCs every 12 months. Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
- Not Randomized - Comparison: Participants in this group fulfilled inclusion criteria into the study but refused participation. These participants were used as comparison to other groups
- Non-Randomized - Reacted to Muffin: At baseline, participants had an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to muffin and were not randomized. Participants were instructed to avoid milk and return for re-evaluation with laboratory tests at 12 and 24 months and baked milk challenge at 36 months
- Non-Randomized - Tolerant to Baked and Non-baked Milk: At baseline, participants had an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group passed all OFCs without a reaction were not randomized. Participants were instructed to include full milk products to their diet for 3 months, followed by complete dietary milk elimination for 1 month. Participants were then re-challenged to unheated milk. Following successful challenge, participants were placed on an unrestricted milk diet and brought in for re-evaluation at 6 months. If participants were not successful in their challenge to unheated milk, they had baked milk products progressively re-introduced to their diets.
Period: Overall Study
Arm/Group | Dose Escalation - Reacted to Pizza | Dose Escalation - Reacted to Rice Pudding | Dose Escalation - Reacted to Non-baked Milk | Maintenance - Reacted to Pizza | Maintenance - Reacted to Rice Pudding | Maintenance- Reacted to Non-baked Milk | Not Randomized - Comparison | Non-Randomized - Reacted to Muffin | Non-Randomized - Tolerant to Baked and Non-baked Milk
Started | 16 | 5 | 20 | 15 | 6 | 23 | 34 | 41 | 10
Completed | 9 | 3 | 10 | 12 | 6 | 13 | 19 | 26 | 6
Not Completed | 7 | 2 | 10 | 3 | 0 | 10 | 15 | 15 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 3 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 8 | 2 | 0 | 6 | 12 | 12 | 4
Not completed — New Contraindication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled
Groups:
- Dose Escalation - Reacted to Rice Pudding: At baseline, participants performed an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to rice pudding and were then randomized to re-try less denatured milk protein food items every 6 months (dose escalation). Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation - Reacted to Pizza | Dose Escalation - Reacted to Rice Pudding | Dose Escalation - Reacted to Non-baked Milk | Maintenance - Reacted to Pizza | Maintenance - Reacted to Rice Pudding | Maintenance- Reacted to Non-baked Milk | Not Randomized - Comparison | Non-Randomized - Reacted to Muffin | Non-Randomized - Tolerant to Baked and Non-baked Milk | Total
Number analyzed (Participants) | 16 | 5 | 20 | 15 | 6 | 23 | 34 | 41 | 10 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (2.3) | 6.2 (1.6) | 7.7 (2.1) | 7.3 (2.2) | 6.7 (2.7) | 6.3 (2.1) | 6.5 (2.3) | 7.5 (1.9) | 6.5 (2.2) | 6.9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 7 | 3 | 3 | 6 | 11 | 12 | 5 | 52
  Male | 12 | 4 | 13 | 12 | 3 | 17 | 23 | 29 | 5 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 5 | 20 | 15 | 6 | 21 | 28 | 38 | 10 | 159
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 3 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 2 | 0 | 3 | 0 | 5 | 1 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  White | 14 | 4 | 18 | 13 | 6 | 18 | 28 | 31 | 9 | 141
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 3 | 0 | 11
Region of Enrollment [Number; unit: participants]
  United States | 16 | 5 | 20 | 15 | 6 | 23 | 34 | 41 | 10 | 170
Baseline Boiled Milk Wheal [Mean (Standard Deviation); unit: Mm] — A skin prick test (SPT) measured the presence of immunoglobulin E (IgE) antibodies for the food tested. During the SPT, a drop of solution containing the food allergen was placed on the forearm. Using a small plastic needle, the skin was gently pricked or scratched to allow a tiny amount of the solution to enter just below the surface. After 15 minutes, positive results were indicated by a wheal, a raised white bump surrounded by a small circle of red skin. The wheal was measured in millimeters. Larger sizes indicated a greater chance of experiencing an allergic reaction to the food tested.
  Mm | 7.3 (2.4) | 6.1 (3.5) | 6.6 (2.8) | 7.6 (1.9) | 7.6 (2.0) | 5.5 (3.2) | 7.7 (4.5) | 7.9 (2.6) | 3.4 (2.5) | 6.9 (3.2)
Baseline Milk Extract Wheal [Mean (Standard Deviation); unit: Mm] — A skin prick test (SPT) measured the presence of immunoglobulin E (IgE) antibodies for the food tested. During the SPT, a drop of solution containing the food allergen was placed on the forearm. Using a small plastic needle, the skin was gently pricked or scratched to allow a tiny amount of the solution to enter just below the surface. After 15 minutes, positive results were indicated by a wheal, a raised white bump surrounded by a small circle of red skin. The wheal was measured in millimeters. Larger sizes indicated a greater chance of experiencing an allergic reaction to the food tested.
  Mm | 8.9 (2.4) | 8.6 (1.2) | 9.1 (3.4) | 8.9 (2.8) | 8.1 (2.7) | 8.5 (3.4) | 9.0 (3.8) | 10.5 (3.7) | 5.0 (2.6) | 8.9 (3.4)
Baseline Unheated Milk Wheal [Mean (Standard Deviation); unit: Mm] — A skin prick test (SPT) measured the presence of immunoglobulin E (IgE) antibodies for the food tested. During the SPT, a drop of solution containing the food allergen was placed on the forearm. Using a small plastic needle, the skin was gently pricked or scratched to allow a tiny amount of the solution to enter just below the surface. After 15 minutes, positive results were indicated by a wheal, a raised white bump surrounded by a small circle of red skin. The wheal was measured in millimeters. Larger sizes indicated a greater chance of experiencing an allergic reaction to the food tested.
  Mm | 10.4 (4.2) | 11.6 (4.2) | 8.3 (2.5) | 8.8 (2.3) | 10.0 (2.7) | 9.7 (4.0) | 9.6 (4.3) | 10.1 (2.6) | 5.6 (2.8) | 9.3 (3.4)
Baseline Cow's Milk IgE [Mean (Standard Deviation); unit: kUa/L] — When cow's milk immunoglobulin E (IgE) antibodies are present in serum samples, this is indicative of a potential for an allergic reaction to cow's milk. The greater the concentration of IgE antibodies present, the more likely an allergic reaction to cow's milk is to occur.
  kUa/L | 10.3 (11.5) | 10.5 (7.8) | 5.3 (5.4) | 7.8 (9.7) | 13.7 (13.1) | 4.1 (4.5) | 14.7 (21.3) | 15.1 (12.7) | 4.9 (8.1) | 10.6 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Progression in Tolerance of Baked Milk and Ultimately Unheated Milk in Dose Escalation Sub-arm Compared to Maintenance Sub-arm
Description: Participants were grouped based on the food to which they experienced a reaction at the baseline Oral Food Challenge (OFC). Group 1=reacted to muffin; Group 2=reacted to pizza; Group 3=reacted to rice pudding; Group 4=reacted to non-baked milk; Group 5=did not react. Groups 2, 3, and 4 were randomized to dose escalation or maintenance, and at each visit following randomization, participants performed an OFC where they were given food products containing milk protein denatured through baking. Participants were given progressively less denatured milk protein food items until they had an allergic reaction. Participants were considered to have a positive progression in tolerance of baked milk if they experienced a reaction to a less denatured milk protein food item at any post randomization visits than the one to which they reacted at their baseline visit.
Time Frame: Randomization through end of study (up to 36 months)
Population: Randomized intent-to-treat
Measure: Number; unit: participants
Groups:
- Dose-Escalation Group: Participants in groups 2-4 were randomized to re-try less denatured milk protein food items every 6 months.
- Maintenance Group: Participants in groups 2-4 were randomized to re-try less denatured milk protein food items every 12 months.
Arm/Group | Dose-Escalation Group | Maintenance Group
Number analyzed (Participants) | 41 | 44
participants | 26 | 31
Statistical Analysis 1: Comparison: Dose-Escalation Group vs Maintenance Group; Test type: Superiority or Other; p = 0.58, Regression, Logistic; Odds Ratio, log = 0.77, 95% CI 2-sided [0.31 to 1.93]

2. Secondary Outcome: Number of Participants With a Positive Progression in Tolerating More Allergenic Forms of Milk at 12 and 24 Months
Description: Participants were grouped based on the food they experienced a reaction to at the baseline Oral Food Challenge (OFC). Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Groups 2, 3 and 4 were randomized to dose escalation or maintenance, and at each visit following randomization, performed an OFC where food products containing milk protein denatured through baking were given. Participants were given progressively less denatured milk protein food items until an allergic reaction occurred. A positive progression in tolerance of baked milk was defined as a reaction to a less denatured milk protein food at 12 months than at baseline. Positive progression at 24 months was defined as experiencing a reaction to a less denatured milk protein food at 24 months than at 12 months.
Time Frame: 12 months, 24 months
Population: Randomized intent-to-treat
Measure: Number; unit: participants
Groups:
- Dose-Escalation Group: Participants in groups 2-4 were randomized to re-try less denatured milk protein food items every 6 months.[Dose Escalation arm].
- Maintenance Group: Participants in groups 2-4 were randomized to re-try less denatured milk protein food items every 12 months.[Maintenance arm].
Arm/Group | Dose-Escalation Group | Maintenance Group
Number analyzed (Participants) | 41 | 44
participants
  Progressed at 12 Months | 18 | 18
  Progressed at 24 Months | 23 | 27
Statistical Analysis 1: Comparison: Dose-Escalation Group vs Maintenance Group; Progression comparison at 12 Months; Test type: Superiority or Other; p = 0.78, Chi-squared; Odds Ratio, log = 1.13, 95% CI 2-sided [0.48 to 2.68]
Statistical Analysis 2: Comparison: Dose-Escalation Group vs Maintenance Group; Progression comparison at 24 Months; Test type: Superiority or Other; p = 0.62, Chi-squared; Odds Ratio, log = 0.81, 95% CI 2-sided [0.34 to 1.91]

3. Secondary Outcome: Percent of Participants Becoming Tolerant to Unheated Cow's Milk at 12, 24, and 36 Months
Description: Participants were grouped based on the food to which they experienced a reaction at the baseline Oral Food Challenge (OFC). Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Groups 2, 3 and 4 were randomized to dose escalation or maintenance, and at each visit following randomization, participants performed an OFC where they were given food products containing milk protein denatured through baking. Participants were given progressively less denatured milk protein food items until they had an allergic reaction. Participants were considered to become tolerant to unheated cow's milk if at the specified visit, they did not react to any of the foods given in the OFC.
Time Frame: 12 months, 24 months, and 36 months
Population: Randomized intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Dose-Escalation Group | Maintenance Group
Number analyzed (Participants) | 41 | 44
percentage of participants
  Tolerant at 12 Month | 29.3 | 15.9
  Tolerant at 24 Months | 43.9 | 29.5
  Tolerant at 36 Months | 53.7 | 43.2
Statistical Analysis 1: Comparison: Dose-Escalation Group vs Maintenance Group; Comparison at 12 Months; Test type: Superiority or Other; p = 0.14, Chi-squared
Statistical Analysis 2: Comparison: Dose-Escalation Group vs Maintenance Group; Comparison at 24 Months; Test type: Superiority or Other; p = 0.17, Chi-squared
Statistical Analysis 3: Comparison: Dose-Escalation Group vs Maintenance Group; Comparison at 36 Months; Test type: Superiority or Other; p = 0.33, Chi-squared

4. Secondary Outcome: Percent of Participants Becoming Tolerant to Unheated Cow's Milk
Description: Participants were grouped based on the food to which they experienced a reaction at the baseline Oral Food Challenge (OFC). Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Groups 2, 3 and 4 were randomized to dose escalation or maintenance, and at each visit following randomization, participants performed an OFC where they were given food products containing milk protein denatured through baking. Participants were given progressively less denatured milk protein food items until they had an allergic reaction. Participants were considered to become tolerant to unheated cow's milk if at any post-randomization visit up through 36 months, they did not react to any of the food given in the OFC.
Time Frame: Randomization through end of study (up to 36 months)
Population: Randomized intent-to-treat
Measure: Number; unit: percentage of participants
Groups:
- Group 2 - Pizza: Participants in this group experienced a reaction to pizza during their baseline visit oral food challenge
- Group 3 - Rice Pudding: Participants in this group experienced a reaction to rice pudding during their baseline visit oral food challenge
- Group 4 - Milk: Participants in this group experienced a reaction to unheated milk during their baseline visit oral food challenge
Arm/Group | Group 2 - Pizza | Group 3 - Rice Pudding | Group 4 - Milk
Number analyzed (Participants) | 31 | 11 | 43
percentage of participants | 38.7 | 54.5 | 53.5
Statistical Analysis 1: Comparison: Group 2 - Pizza vs Group 3 - Rice Pudding vs Group 4 - Milk; Test type: Superiority or Other; p = 0.41, Chi-squared

5. Secondary Outcome: Comparison of Baseline Basophil Percent Maximal Degranulation With the Outcome of the Baseline OFC to Identify the Biomarkers of Clinical Reactivity
Description: This endpoint evaluates the correlation between the mechanistic biomarkers of basophil reactivity and the food to which participants reacted at baseline. Participants were grouped according to food at which participants experienced a reaction during their baseline oral food challenge: Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Basophils come from blood drawn at baseline. Basophils counts were done using whole blood specimens. Basophil reactivity as measured as maximal degranulation percentage after stimulation with titrated dilutions of milk powder (from 1x103 to 1x10-1 µg/mL total protein) and was correlated to group assignment using Spearman correlation coefficients.
Time Frame: Baseline
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: percentage of max basophil degranulation
Groups:
- Group 1 = Muffin: Participants in this group experienced an allergic reaction to eating a muffin during their baseline oral food challenge
- Group 2 = Pizza: Participants in this group experienced an allergic reaction to eating pizza during their baseline oral food challenge
- Group 3 = Rice Pudding: Participants in this group experienced an allergic reaction to eating rice pudding during their baseline oral food challenge
- Group 4 = Milk: Participants in this group experienced an allergic reaction to drinking unheated milk during their baseline oral food challenge
- Group 5 = Passed All: Participants in this group passed all oral food challenges without an allergic reaction during their baseline visit
Arm/Group | Group 1 = Muffin | Group 2 = Pizza | Group 3 = Rice Pudding | Group 4 = Milk | Group 5 = Passed All
Number analyzed (Participants) | 41 | 31 | 11 | 43 | 10
percentage of max basophil degranulation | 41.0 [16.9 to 76.7] | 29.3 [12.8 to 47.8] | 45.6 [13.9 to 85.3] | 20.3 [6.3 to 55.1] | 8.9 [6.7 to 32.1]
Statistical Analysis 1: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Test type: Superiority or Other; p = 0.09, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Test type: Superiority or Other; p = 0.01, Spearman's Correlation — Null hypothesis is that correlation = 0

6. Secondary Outcome: Comparison of Baseline IgE With the Outcome of the Baseline OFC to Identify the Biomarkers of Clinical Reactivity
Description: This endpoint evaluates the correlation between the mechanistic biomarker of IgE to milk proteins and allergic reaction at baseline. Participants were grouped according to food at which participants experienced a reaction during their baseline oral food challenge: Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Quantitative IgE to milk proteins was done using FEIA (UniCAP) on serum from blood drawn at baseline.
Time Frame: Baseline
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: kUa/L
Arm/Group | Group 1 = Muffin | Group 2 = Pizza | Group 3 = Rice Pudding | Group 4 = Milk | Group 5 = Passed All
Number analyzed (Participants) | 41 | 31 | 11 | 43 | 10
kUa/L
  Beta-lactoglobulin IgE | 1.9 [0.6 to 4.0] | 0.6 [0.2 to 2.4] | 1.3 [0.4 to 3.5] | 0.4 [0.2 to 2.3] | 0.2 [0.2 to 0.4]
  Casein IgE | 12.3 [3.4 to 17.9] | 4.1 [1.6 to 9.6] | 5.6 [2.0 to 12.9] | 1.6 [0.7 to 3.6] | 0.8 [0.2 to 1.6]
  Cow's Milk IgE | 12.1 [5.0 to 21.1] | 5.4 [2.1 to 12.2] | 7.7 [3.9 to 19.1] | 3.5 [1.7 to 5.6] | 0.9 [0.2 to 4.3]
Statistical Analysis 1: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Betalactoglobulin; Test type: Superiority or Other; p < 0.01, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Betalactoglobulin IgE; Test type: Superiority or Other; p < 0.01, Spearman Correlation — Null hypothesis is that correlation = 0
Statistical Analysis 3: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Casein IgE; Test type: Superiority or Other; p < 0.01, Kruskal-Wallis
Statistical Analysis 4: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Casein IgE; Test type: Superiority or Other; p < 0.01, Spearman Correlation — Null hypothesis is that correlation = 0
Statistical Analysis 5: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Cow's Milk IgE; Test type: Superiority or Other; p < 0.01, Kruskal-Wallis
Statistical Analysis 6: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Cow's Milk IgE; Test type: Superiority or Other; p < 0.01, Spearman Correlation — Null hypothesis is that correlation = 0

7. Secondary Outcome: Comparison of Baseline Mechanistic Studies [Treg and Basophil] With the Outcome of the Baseline OFC to Identify the Biomarkers of Clinical Reactivity
Description: This endpoint evaluates the correlation between the mechanistic biomarker of the number of basophils and T regulatory cells reactive to milk proteins and the food to which participants reacted at baseline. Participants were grouped according to food at which participants experienced a reaction during their baseline oral food challenge: Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Quantitative IgE to milk proteins was done using FEIA (UniCAP) on serum from blood drawn at baseline.
Time Frame: Baseline
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Group 1 = Muffin | Group 2 = Pizza | Group 3 = Rice Pudding | Group 4 = Milk | Group 5 = Passed All
Number analyzed (Participants) | 41 | 31 | 11 | 43 | 10
cells/µL
  Max Basophil Assessment | 1160.0 [635.0 to 1981.0] | 717.0 [456.0 to 982.0] | 1589.5 [1287.5 to 3972.0] | 934.0 [459.0 to 1669.0] | 524.0 [319.0 to 1087.0]
  Tregs | 4.2 [2.4 to 7.0] | 6.2 [2.4 to 8.5] | 7.5 [2.4 to 12.5] | 5.2 [3.5 to 10.1] | 4.2 [2.2 to 8.5]
Statistical Analysis 1: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Max Basophil Assessment; Test type: Superiority or Other; p = 0.01, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Max Basophil Assessment; Test type: Superiority or Other; p = 0.22, Spearman Correlation — Null hypothesis is that correlation = 0
Statistical Analysis 3: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Tregs; Test type: Superiority or Other; p = 0.59, Kruskal-Wallis
Statistical Analysis 4: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Analysis on Tregs; Test type: Superiority or Other; p = 0.32, Spearman Correlation — Null hypothesis is that correlation = 0

8. Secondary Outcome: Relationship Between Initial Dose of Tolerated Baked-milk Protein and Time to Complete Tolerance
Description: Participants were grouped based on the food to which they experienced a reaction at the baseline Oral Food Challenge (OFC). Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Groups 2, 3 and 4 were randomized to dose escalation or maintenance, and at each visit following randomization, participants performed an OFC where they were given food products containing milk protein denatured through baking. Participants were given progressively less denatured milk protein food items until they had an allergic reaction. Participants were considered to become tolerant to unheated cow's milk if at any post-randomization visit up through 36 months, they did not react to any food, including unheated whole milk.
Time Frame: Randomization through end of study (up to 36 months)
Population: Randomized intent-to-treat participants who achieved tolerance
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Group 2 - Pizza | Group 3 - Rice Pudding | Group 4 - Milk
Number analyzed (Participants) | 12 | 6 | 23
months | 24.0 (12.6) | 17.8 (12.7) | 19.6 (10.7)
Statistical Analysis 1: Comparison: Group 2 - Pizza vs Group 3 - Rice Pudding vs Group 4 - Milk; Test type: Superiority or Other; p = 0.50, Kruskal-Wallis

9. Secondary Outcome: Relationship Between Dose of Baked-milk Protein and Reactivity to Casein Versus Whey
Description: Participants were grouped based on the food to which they experienced a reaction at the baseline Oral Food Challenge (OFC). Group 1 = reacted to muffin; Group 2 = reacted to pizza; Group 3 = reacted to rice pudding; Group 4 = reacted to non-baked milk; Group 5 = did not react. Groups 2, 3 and 4 were randomized to dose escalation or maintenance, and at each visit following randomization, participants performed an OFC where they were given food products containing milk protein denatured through baking. Participants were given progressively less denatured milk protein food items until they had an allergic reaction. The relationship between serum IgE to betalactoglobulin and casein, and the food level at which the participant reacted, were evaluated at each post randomization OFC visit. It is expected that those who reacted to muffin would have a higher ratio of casein to betalactoglobulin than those who reacted to less heated forms of milk.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Group 1 = Muffin | Group 2 = Pizza | Group 3 = Rice Pudding | Group 4 = Milk | Group 5 = Passed All
Number analyzed (Participants) | 41 | 31 | 11 | 43 | 10
Ratio
  Baseline | 4.6 [3.0 to 6.5] | 4.6 [1.8 to 9.0] | 5.5 [0.9 to 14.2] | 2.1 [1.0 to 6.6] | 1.6 [1.0 to 9.4]
  Month 12 Visit | 7.7 [4.7 to 20.7] | 3.0 [2.0 to 12.2] | 4.5 [3.1 to 11.5] | 2.3 [1.1 to 4.3] | 2.2 [1.0 to 7.0]
  Month 24 Visit | 3.7 [1.4 to 7.6] | 3.3 [3.0 to 9.2] | 4.8 [2.8 to 171.2] | 1.0 [0.9 to 6.2] | 2.6 [1.0 to 3.7]
  Month 36 Visit | 4.6 [2.5 to 9.0] | 2.5 [2.1 to 13.7] | 5.1 [0.4 to 6.2] | 1.1 [1.0 to 2.6] | 2.3 [1.0 to 27.3]
Statistical Analysis 1: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Baseline Comparison; Test type: Superiority or Other; p = 0.033, Spearman Correlation — Correlation = -0.18
Statistical Analysis 2: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Month 12 Comparison; Test type: Superiority or Other; p = 0.002, Spearman Correlation — Correlation = -0.34
Statistical Analysis 3: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Month 24 Comparison; Test type: Superiority or Other; p = 0.156, Spearman Correlation — Correlation = -0.20
Statistical Analysis 4: Comparison: Group 1 = Muffin vs Group 2 = Pizza vs Group 3 = Rice Pudding vs Group 4 = Milk vs Group 5 = Passed All; Month 36 Comparison; Test type: Superiority or Other; p = 0.077, Spearman Correlation — Correlation = -0.27

10. Secondary Outcome: Comparison of Percent of Participants Tolerant to Non-heated Milk Between the Participants Who Ingested Baked-milk Products and Participants Who Continued to Avoid All Forms of Milk
Description: Participants were grouped based on the food they reacted to, at the baseline Oral Food Challenge (OFC). Group 1= reacted to muffin; Group 2= reacted to pizza; Group 3= reacted to rice pudding; Group 4= reacted to non-baked milk; Group 5= did not react. Groups 2- 4 were randomized to dose escalation or maintenance, and Group 1, and a Control group that chose not to participate in the study, continued to avoid milk. Randomized participants performed an OFC at each visit during which they were given progressively less denatured/ baked milk protein food items until they had an allergic reaction. Participants were considered tolerant to unheated cow's milk if at any post-randomization visit up through 36 months, they did not react to any food, including unheated whole milk. Tolerance of non-heated milk was assessed by report among those who continued to avoid milk.
Time Frame: Month 36
Population: Randomized and comparison participants
Measure: Number; unit: percent participants
Groups:
- Active: This group included participants who were in baseline groups 2 through 4.
- Comparison Group: This group comprised of participants who did not want to participate in OFCs and were advised to avoid milk-based food products for the remainder of the study
- Reacted to Muffin: This group included participants who were in baseline group 1
Arm/Group | Active | Comparison Group | Reacted to Muffin
Number analyzed (Participants) | 85 | 34 | 41
percent participants | 48.2 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Active vs Comparison Group vs Reacted to Muffin; 36 Month Comparison; Test type: Superiority or Other; p < 0.01, Chi-squared

11. Secondary Outcome: Changes in Mechanistic Values [Humoral, T Cell and Basophil]
Description: This outcome measure was not well defined in the protocol and was not analyzed.
Time Frame: Baseline, Month 12, Month 24, and Month 36
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Active | Comparison Group | Reacted to Muffin
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Changes in Mechanistic Values [Humoral, T Cell and Basophil]
Description: This outcome measure was not well defined in the protocol and was not analyzed.
Time Frame: Baseline to the time complete milk tolerance was established
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Active | Comparison Group | Reacted to Muffin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment through end of study (up to 3 years)
Groups:
- Maintenance - Reacted to Non-baked Milk: At baseline, participants had an oral food challenge (OFC). They were given food containing milk protein denatured through baking. Participants were given progressively increasing quantities of less denatured milk protein foods until they had an allergic reaction. The food they experienced a reaction to was their baseline group. Participants in this group reacted to rice pudding and were then randomized to continue eating the food at the same level of milk denaturalization and come in for OFCs every 12 months. Participants in this group received instructions for intake of baked milk foods at home and were followed up to 46 months.
Arm/Group | Dose Escalation - Reacted to Pizza | Dose Escalation - Reacted to Rice Pudding | Dose Escalation - Reacted to Non-baked Milk | Maintenance - Reacted to Pizza | Maintenance - Reacted to Rice Pudding | Maintenance - Reacted to Non-baked Milk | Not Randomized - Comparison | Non-Randomized - Reacted to Muffin | Non-Randomized - Tolerant to Baked and Non-baked Milk
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/5 | 0/20 | 0/15 | 1/6 | 0/23 | 0/34 | 0/41 | 0/10
Other Adverse Events (participants affected / at risk) | 16/16 | 5/5 | 20/20 | 15/15 | 6/6 | 23/23 | 20/34 | 40/41 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation - Reacted to Pizza (N=16) | Dose Escalation - Reacted to Rice Pudding (N=5) | Dose Escalation - Reacted to Non-baked Milk (N=20) | Maintenance - Reacted to Pizza (N=15) | Maintenance - Reacted to Rice Pudding (N=6) | Maintenance - Reacted to Non-baked Milk (N=23) | Not Randomized - Comparison (N=34) | Non-Randomized - Reacted to Muffin (N=41) | Non-Randomized - Tolerant to Baked and Non-baked Milk (N=10)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation - Reacted to Pizza (N=16) | Dose Escalation - Reacted to Rice Pudding (N=5) | Dose Escalation - Reacted to Non-baked Milk (N=20) | Maintenance - Reacted to Pizza (N=15) | Maintenance - Reacted to Rice Pudding (N=6) | Maintenance - Reacted to Non-baked Milk (N=23) | Not Randomized - Comparison (N=34) | Non-Randomized - Reacted to Muffin (N=41) | Non-Randomized - Tolerant to Baked and Non-baked Milk (N=10)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Growth hormone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Food allergy (Immune system disorders) | 15 (53) | 4 (7) | 13 (31) | 14 (66) | 6 (19) | 16 (48) | 13 (18) | 39 (104) | 2 (11)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 9 (18) | 3 (4) | 18 (40) | 12 (24) | 5 (12) | 23 (49) | 5 (6) | 14 (19) | 1 (8)
Seasonal allergy (Immune system disorders) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (3) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 3 (5) | 2 (2) | 4 (5) | 1 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 3 (4) | 4 (6) | 3 (6) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 5 (7) | 3 (4) | 4 (5) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 4 (5) | 4 (7) | 3 (4) | 2 (4) | 1 (1) | 4 (5) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No